CLINICAL TRIAL: NCT05718388
Title: Effect of Contralateral Isokinetic Training on Strength and Reaching Skill in Children With Spastic Hemiplegic Cerebral Palsy
Brief Title: Contralateral Isokinetic Training on Strength and Reaching Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant professor at faculty of physical therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: contralateral isokinetic
Record Dates: First submitted 2023-01-21; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hemiplegic Cerebral Palsy
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (A) (Other): They received a physiotherapy program
  Interventions: Other: Physical therapy exercises
- study Group (B) (Experimental): They received the same program given to control group (A) in addition to isokinetic resistance training of the less affected upper limb for shoulder abductors in concentric mode at the angular velocity of 180 degree/ second
  Interventions: Other: Isokinetic training

INTERVENTIONS:
Other: Physical therapy exercises — For two consecutive months, the children in control group underwent a physiotherapy program for 60min/ three sessions each week: it was based mainly on the neurodevelopment technique, directed toward inhibiting abnormal muscle tone facilitating normal patterns of postural control and hand functions training program
  Arms: Control group (A)
Other: Isokinetic training — Children in study group received the same program given to control group (A) in addition to isokinetic resistance training of the less affected upper limb for shoulder abductors in concentric mode at the angular velocity of 180 degree/ second under full supervision on the Biodex isokinetic dynamometer three times per week for 8 weeks, making a total of 24 training sessions. Each child was trained in the seated position with the similar precaution of the testing protocol.
  Arms: study Group (B)

SUMMARY:
The study aimed to ascertain how cross-education affected the activity of the paretic muscles in the upper limb and how that affected function in children with spastic hemiplegia and cerebral palsy. Additionally, it sought to determine how unilateral isokinetic resistance training affected children with spastic hemiplegia of the contralateral limb in terms of strength development.

ELIGIBILITY:
Inclusion Criteria:

* hemiplegic CP children from both genders with age ranged from five to seven year
* had mild to moderate spasticity according to the Modified Ashworth Scale
* able to follow verbal instructions
* able to stand unassisted and ambulate with abnormal pattern

Exclusion Criteria:

* children who had any visual or auditory problems, fixed deformities in upper limb that interfere with fine motor functions, with history of any surgical interference in upper limbs for less than one year, and un-cooperative children were excluded.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Concentric isokinetic shoulder abductors peak torque in Newton- meters and average power. | Change from Baseline Isokinetic dynamometer parameters at 2 months
  Isokinetic dynamometer was used to measure the concentric isokinetic shoulder abductors peak torque in Newton- meters and average power at an angular velocity of 180 degrees per second in concentric mode with gravity adjustment

SECONDARY OUTCOMES:
Modified functional scale for reaching | Change from Baseline Modified functional scale for reaching at 2 months
  It was used to measure the ability of the child to perform the reaching skills. It was used to determine the level of performance and functional improvement in reaching skills. Each child was seated in front of a table, in a chair adjustable to his or her height. They were appropriately fitted and supported to avoid any substitution movement from the child's trunk. The target was positioned on the top of the table, beside the child. The child's elbow was passively placed at full extension and the writ in natural position. Each trail of the reaching task was begun with the child's arm straight and parallel to the patient's trunk. The child was asked to make accurate reaching to touch the target by the affected arm when the examiner gives the command.

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No